CLINICAL TRIAL: NCT06640595
Title: Simulation Study on Advanced Medical Procedures Under Extreme Environments
Acronym: SIMEX-MED
Status: Completed | Type: Observational
Sponsor: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Principal Investigator, Simon Rauch, Senior Researcher, Institute of Mountain Emergency Medicine
Other Study IDs: SIMEX-MED
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Cold Exposure
Keywords: Intubation; Front of neck access; Mini-Thoracotomy; Cold temperature

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cold Temperature: Performance of the procedure under cold temperature (-20°C)
- Normal Temperature: Performance of the procedure under normal temperature (+20°C)

SUMMARY:
Background:

In emergency situations in mountainous regions, medical professionals are often required to perform advanced medical procedures swiftly and efficiently. The choice of procedure and the environmental conditions can significantly impact the patient outcomes. This study seeks to evaluate the effectiveness of three advanced emergency medical procedures in a simulated scenario: orotracheal intubation with a videolaryngoscopy, minithoracotomy, and front of neck access, under both normal and cold temperature conditions.

Methods:

On 16 and 17 October 2023, members of the Medical Commission of the International Commission for Alpine Rescue performed a simulation training in an extreme environmental simulation chamber (terraXcube) in Bolzano, Italy. During this, each participant will perform three advanced medical procedures, once under normal environmental conditions (+20°C) and once under cold temperature conditions (-20°C), in randomized order and with a crossover design. Specifically, the three advanced medical procedures consist of 1) simulation of a difficult orotracheal intubation on a dedicated mannikin with a videolaryngoscope; 2) front of neck access (FONA) with the scalpel-finger-bougie technique on a dedicated mannikin model; 3) minithoracotomy and chest tube placement on a dedicated mannikin model.

Outcomes:

Primary outcome:

The primary outcome is the difference in time required for three different advanced medical procedures, i.e. orotracheal intubation with a videolaryngoscopy, minithoracotomy, and front of neck access, under normal environmental conditions (+20°C) compared to cold temperature (-20°C).

Secondary outcomes:

Secondary outcomes include the success rate for three different advanced medical procedures, i.e. orotracheal intubation with a videolaryngoscopy, minithoracotomy, and front of neck access, under normal environmental conditions (+20°C) compared to cold temperature (-20°C). Moreover, the subjective difficulty of performing the procedures, stress levels, emotional regualtion and decision-making process will be assessed through a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Members of the Medical Commission of the International Commission for Alpine Rescue (ICAR)

Exclusion Criteria:

* Contraindications for exposure to cold temperatures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of the Medical Commission of the International Commission for Alpine Rescue (ICAR)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Difference in Time to perform the procedure | During the performance of the procedure
  Difference in time required to perform three different advanced medical procedures, i.e. orotracheal intubation with a videolaryngoscopy, minithoracotomy, and front of neck access, under normal environmental conditions (+20°C) compared to cold temperature (-20°C).

SECONDARY OUTCOMES:
Success rate | During the procedure
  Success rate for three different advanced medical procedures, i.e. orotracheal intubation with a videolaryngoscopy, minithoracotomy, and front of neck access, under normal environmental conditions (+20°C) compared to cold temperature (-20°C).
Stress level | Immediately after the performance of the procedure
  Stress levels of the participants will be assessed through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rauch, MD, PhD, Principal Investigator — Institute of Mountain Emergency Medicine, Eurac research
Locations (1):
- Eurac Research, Bolzano, Italy

IPD SHARING:
Plan to Share IPD: No